CLINICAL TRIAL: NCT03507894
Title: Impact of M-health Based Intervention on Adherence to Healthy Physical Activity After Stroke. Randomized Study
Brief Title: Impact of M-health Based Intervention on Adherence to Healthy Physical Activity After Stroke.
Status: Completed | Type: Observational
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Montserrat Grau-Pellicer, Principal Investigator, Consorci Sanitari de Terrassa
Other Study IDs: ConsorciST
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Stroke
Keywords: rehabilitation; exercise; stroke; adherence
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- m-health stroke rehabilitation: 8-week multimodal exercise rehabilitation program (MERP) based on aerobic exercise, task oriented activities, balance and stretching exercises complemented with a mobile app technology
  Interventions: Behavioral: Multimodal Exercise Rehabilitation Program

INTERVENTIONS:
Behavioral: Multimodal Exercise Rehabilitation Program — Rehabilitation program based on aerobic exercise, task oriented activities, balance and stretching exercises complemented with a mobile app technology

SUMMARY:
The aim of this study is to determine the impact of an m-health based intervention on long term adherence to a rehabilitation program for stroke survivors.

DETAILED DESCRIPTION:
This is a 8-week multimodal exercise rehabilitation program (MERP) based on aerobic exercise, task oriented activities, balance and stretching exercises complemented with a mobile app technology. The aim of the MERP is to improve walking speed, walking ability, activities of daily living and quality of life among people who have suffered a stroke. The mobile app technology complements the MERP in order to achieve long term adherence to healthy physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic or hemorrhagic stroke
* age ≥18;
* Functional Ambulation Classification (FAC) ≥3
* Barthel Index ≥45

Exclusion Criteria:

* Cognitive impairment (Mini Mental State Examination ≤24)
* Unstable cardiovascular disease (acute heart failure, recent myocardial infarction, unstable angina and uncontrolled arrhythmias)
* Alcohol or other toxic substances abuse
* Decompensated psychiatric disorders that prevented from following a group session

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be stroke survivors who have completed a conventional rehabilitation program. They will be recruited from Hospital-Consorci Sanitari de Terrassa (Barcelona, Spain) over a period of six months.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Adherence | 8 weeks
  Adherence will be monitored with an app that will record activity time (walking time and distance)

SECONDARY OUTCOMES:
Gait speed | 8 weeks
  Gait speed will be measured with the Ten Meter Walking Test (10MWT). Participants will be given a 2-meter warm-up distance for walking, preceding the 10-meter distance, and 2 meters beyond the 10 meters. The time that takes to walk 10 meters at a comfortable pace and at their maximum speed will be registered in meters/second

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Grau-Pellicer, PhD, Principal Investigator — Consorci Sanitari de Terrassa
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saunders DH, Mead GE, Fitzsimons C, Kelly P, van Wijck F, Verschuren O, Backx K, English C. Interventions for reducing sedentary behaviour in people with stroke. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD012996. doi: 10.1002/14651858.CD012996.pub2. PMID 34184251